CLINICAL TRIAL: NCT06375902
Title: The Fragility of Metaphors (FraMe): Learning, Loosing, and How to Train Them
Acronym: FRAME
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marta Bosia, Prof.ssa, IRCCS San Raffaele
Other Study IDs: 2022289RNA
Record Dates: First submitted 2024-03-15; First posted 2024-04-19 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; Psychosis
Keywords: language; pragmatics; rehabilitation; electrophysiology
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Schizophrenia group: We will enroll 32 patients selected according to the presence of Schizophrenia diagnosis (DSM V criteria), which will be tested for metaphor comprehension, as well as for the other variables included in the study, and the electrical brain activity will be registered through a 128 channel EEG.
  Patients will be assigned either to a rehabilitative training (PragmaCom), or to a standard rehabilitative program to test if the altered neurophysiological patterns associated to the fragility of metaphor comprehension in schizophrenia can be restored.
  Interventions: Behavioral: PragmaCom
- Healthy controls group: 32 healthy subjects, as control sample, that will be tested for metaphor comprehension, as well as for the other variables included in the study, and the electrical brain activity will be registered through a 128 channel EEG.

INTERVENTIONS:
Behavioral: PragmaCom — Cognitive behavioral intervention targeting the ability to understand metaphors
  Groups: Schizophrenia group

SUMMARY:
Tracking down the difficulties in metaphor comprehension experienced by individuals with schizophrenia across different metaphor types and exploring the neurological correlates via EEG recording technique

DETAILED DESCRIPTION:
The investigators will address the following objectives:

* Primary Objective: Tracking down the difficulties in metaphor comprehension experienced by individuals with schizophrenia across different metaphor types and exploring the neurological correlates via EEG recording technique
* Secondary Objectives: 1) Evaluate the interactions between performances in metaphor comprehension and individual differences in psychopathology, cognition, ToM and functioning; 2) Test if the altered neurophysiological patterns associated to the fragility of metaphor comprehension in schizophrenia can be restored through a rehabilitative training

The investigators will enroll 32 schizophrenic patients and 32 healthy subjects as control sample.

Participants will undergo an initial visit with a specialist psychiatrist who will verify that their conditions meet the criteria required by the study. Then, subjects will be tested for metaphor comprehension, as well as for the other variables included in the study, and the electrical brain activity will be registered through a 128 channel EEG.

In the check-up visits (i.e., after the training) the following data will be collected:

* Scores relating to cognitive, pragmatic (understanding of metaphors), theory of mind and global functioning performance scores
* EEG recordings related to the process of understanding metaphors
* Scores on scales that evaluate psychopathological severity

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Age between 18 and 65 years
* Diagnosis of Schizophrenia according to DSM V criteria
* Ability to provide informed consent

For healthy controls:

* Age between 18 and 65 years
* Ability to provide informed consent
* Absence of psychiatric pathologies
* Ability to speak Italian

Exclusion Criteria:

For patients:

* Intellectual disability
* Neurological disorder

For healthy controls:

* Presence of psychiatric pathologies
* Difficulties in speaking Italian

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 32 Schizophrenic patients and 32 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Tracking down the difficulties in metaphor comprehension via a behavioural task | through study completion, an average of 2 years
  Tracking down the difficulties in metaphor comprehension experienced by individuals with schizophrenia compared to healthy controls across different metaphor types through the Physical and mental metaphor task (PMM) (range values 0-28, higher scores mean a better outcome).
Tracking down the difficulties in metaphor comprehension via task during electrophysiological recording | through study completion, an average of 2 years
  Exploring the difference in the neurological correlates (via electrophysiological recording technique) between patients and controls. Electrophysiological indexes that will be evaluated are event-related potential after the stimulus presentation.

SECONDARY OUTCOMES:
Evaluation of psychopathology | through study completion, an average of 2 years
  Evaluate psychopathology with the Positive and Negative Syndrome scale (PANSS) (range values 30-210, higher scores mean a worse outcome).
Evaluation of cognition | through study completion, an average of 2 years
  Evaluate cognition in schizophrenia with the Brief assessement of cognition in schizophrenia (BACS) (range total score 0-1, higher scores mean a better outcome).
Evaluation of Theory of Mind | through study completion, an average of 2 years
  Evaluate Theory of Mind with the Picture sequencing task (PST) (range score 0-56, higher scores mean a better outcome).
Evaluation of functioning | through study completion, an average of 2 years
  Evaluate functioning, with the Quality of life scale (QLS) (range score 0-126, higher scores mean a better outcome).
Evaluate the efficacy of a rehabilitative training in restoring metaphor comprehension ability | through study completion, an average of 2 years
  Test te improvement of metaphor comprehension, evaluated with the Physical and mental metaphor task (PMM) (range values 0-28, higher scores mean a better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Mart Bosia, MD, PhD, Principal Investigator — Vita-Salute San Raffaele University
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bambini V, Agostoni G, Buonocore M, Tonini E, Bechi M, Ferri I, Sapienza J, Martini F, Cuoco F, Cocchi F, Bischetti L, Cavallaro R, Bosia M. It is time to address language disorders in schizophrenia: A RCT on the efficacy of a novel training targeting the pragmatics of communication (PragmaCom). J Commun Disord. 2022 May-Jun;97:106196. doi: 10.1016/j.jcomdis.2022.106196. Epub 2022 Feb 2. PMID 35526293
- [Background] Thoma P, Daum I. Neurocognitive mechanisms of figurative language processing--evidence from clinical dysfunctions. Neurosci Biobehav Rev. 2006;30(8):1182-205. doi: 10.1016/j.neubiorev.2006.09.001. Epub 2006 Oct 31. PMID 17079014
- [Background] Harvey PD, Bowie CR, Friedman JI. Cognition in schizophrenia. Curr Psychiatry Rep. 2001 Oct;3(5):423-8. doi: 10.1007/s11920-996-0038-7. PMID 11559481
- [Background] Rossetti I, Brambilla P, Papagno C. Metaphor Comprehension in Schizophrenic Patients. Front Psychol. 2018 May 9;9:670. doi: 10.3389/fpsyg.2018.00670. eCollection 2018. PMID 29867648
- [Background] Rapp AM, Felsenheimer AK, Langohr K, Klupp M. The Comprehension of Familiar and Novel Metaphoric Meanings in Schizophrenia: A Pilot Study. Front Psychol. 2018 Jan 5;8:2251. doi: 10.3389/fpsyg.2017.02251. eCollection 2017. PMID 29354082
- [Background] Bambini V, Arcara G, Bosinelli F, Buonocore M, Bechi M, Cavallaro R, Bosia M. A leopard cannot change its spots: A novel pragmatic account of concretism in schizophrenia. Neuropsychologia. 2020 Mar 2;139:107332. doi: 10.1016/j.neuropsychologia.2020.107332. Epub 2020 Jan 7. PMID 31923528
- [Background] Mossaheb N, Aschauer HN, Stoettner S, Schmoeger M, Pils N, Raab M, Willinger U. Comprehension of metaphors in patients with schizophrenia-spectrum disorders. Compr Psychiatry. 2014 May;55(4):928-37. doi: 10.1016/j.comppsych.2013.12.021. Epub 2014 Jan 14. PMID 24556517
- [Background] Bambini V, Bertini C, Schaeken W, Stella A, Di Russo F. Disentangling Metaphor from Context: An ERP Study. Front Psychol. 2016 May 3;7:559. doi: 10.3389/fpsyg.2016.00559. eCollection 2016. PMID 27199799
- [Background] De Grauwe S, Swain A, Holcomb PJ, Ditman T, Kuperberg GR. Electrophysiological insights into the processing of nominal metaphors. Neuropsychologia. 2010 Jun;48(7):1965-84. doi: 10.1016/j.neuropsychologia.2010.03.017. Epub 2010 Mar 20. PMID 20307557
- [Background] Iakimova G, Passerieux C, Laurent JP, Hardy-Bayle MC. ERPs of metaphoric, literal, and incongruous semantic processing in schizophrenia. Psychophysiology. 2005 Jul;42(4):380-90. doi: 10.1111/j.1469-8986.2005.00303.x. PMID 16008767
- [Background] Adamczyk P, Jani M, Ligeza TS, Plonka O, Bladzinski P, Wyczesany M. On the Role of Bilateral Brain Hypofunction and Abnormal Lateralization of Cortical Information Flow as Neural Underpinnings of Conventional Metaphor Processing Impairment in Schizophrenia: An fMRI and EEG Study. Brain Topogr. 2021 Jul;34(4):537-554. doi: 10.1007/s10548-021-00849-x. Epub 2021 May 10. PMID 33973137
- [Background] Bambini V, Tonini E, Ceccato I, Lecce S, Marocchini E, Cavallini E. How to improve social communication in aging: Pragmatic and cognitive interventions. Brain Lang. 2020 Dec;211:104864. doi: 10.1016/j.bandl.2020.104864. Epub 2020 Nov 1. PMID 33137591